CLINICAL TRIAL: NCT05958446
Title: Home Monitoring of Fetal Heart Rhythm in Pregnancies of Anti-Ro/SSA Positive Women for the Treatment of Congenital Heart Block (FETAL HOPE)
Brief Title: Fetal-Hope Study: Home Monitoring of Fetal Heart Rate in SSA+ Pregnant Women
Acronym: FH
Status: Recruiting | Type: Observational
Sponsor: ASST Fatebenefratelli Sacco (Other)
Responsible Party: Principal Investigator, Dr Emanuele Bizzi, Medical Doctor, ASST Fatebenefratelli Sacco
Other Study IDs: 2021/ST/247
Record Dates: First submitted 2023-06-30; First posted 2023-07-24 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Pregnancy Related; Autoimmune Diseases; Neonatal Lupus; SLE; Sjogren's Syndrome; Fetal Heart Rate or Rhythm Abnormality Affecting Fetus
Keywords: sjogren's syndrome; SSA; SLE; pregnancy; fetal heart rate; neonatal lupus
MeSH Terms: conditions — Autoimmune Diseases; Neonatal Systemic lupus erythematosus; Sjogren's Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant women with SSA Auto Ab: All patients over the age of 18, who will sign the informed consent for participation in the study, characterized by the positivity of autoantibodies against Ro/SSA who will become pregnant during the enrollment period.

SUMMARY:
Serological positivity for anti Ro-SSA antibodies is frequently found in pathologies such as Sjogren's Syndrome and SLE. Worldwide, approximately 0.5-1% of women of reproductive age are positive for Ro-SSA antibodies, and in 1-2% of these women, pregnancy will be complicated by cardiac abnormalities of the fetus, particularly varying degrees of atrioventricular block. It is essential to promptly identify patients with fetal heart rhythm abnormalities to prevent both intrauterine deaths and the birth of newborns with third-degree atrioventricular block, requiring lifelong cardiac pacing. At the moment, the only means to identify these alterations is represented by fetal cardiac ultrasound. Fetal atrioventricular block can develop within a few hours in these patients and fetal ultrasound, normally performed no more frequently than once every two weeks, does not allow for the timely identification of these conditions and therefore for pharmacological intervention.

Using home fetal heart rate monitoring, carried out directly by patients three times a day with the aid of a special device that allows easy identification of the fetal heart rhythm, would allow rapid recognition of rhythm alterations and early access to confirmation tests and possible therapies.

Fetal heart rhythm surveillance could detect a medically reversible disease that, if untreated, would progress to lifelong cardiac pacing, with its many associated comorbidities. Applying such protocol in pregnant women anti-Ro/SSA positive could become standard practice.

The main objectives of this study are:

* Estimation of the incidence of the development of fetal AV conduction abnormalities in patients with positivity for Ro/SSA autoantibodies;
* Estimation of the reliability of home monitoring of fetal heart rate with fetal Doppler device in detecting fetal atrioventricular conduction disturbances;
* Evaluation of the results of the therapy administered early, immediately after the diagnosis of fetal atrioventricular conduction disorders.

DETAILED DESCRIPTION:
The association between the transplacental passage of maternal autoantibodies against antigen A (Ro /SSA), common in autoimmune diseases such as Sjögren syndrome (SS) and systemic lupus erythematosus (SLE), and congenital heart block (CHB) has been established for some time.

Worldwide, approximately 0.5-1% of women of reproductive age are positive for anti-Ro/SSA antibodies, and in 1-2% of these women, pregnancy will be complicated by cardiac abnormalities of the fetus, particularly atrioventricular blocks (AVB) of various degrees.

Complete third-degree AVB occurs in 2-4% of fetuses exposed to anti-Ro/SSA, but up to one-third of cases show transient signs of first-degree AVB. Fetal irreversible complete AVB related to maternal Ro/SSA autoantibodies typically develops between weeks 20 and 24 of gestation. This condition has a mortality rate of 17-30%, is burdened by heavy cardiac pacing morbidity throughout the life of children born with AVB, and a high (10 times greater) risk of recurrence in subsequent pregnancies.

Some cases with CHB are preceded by first or second degree heart block. Treatment with steroids has also been suggested to prevent progression of first or second degree heart block to CHB, although the effect is controversial.

Complete or third-degree AVB appears to be irreversible, but anecdotal reports suggest that treatment of second-degree AVB can restore sinus rhythm. Unfortunately, weekly or biweekly fetal echocardiographic surveillance has only rarely detected AVB in time for treatment to be successful.

One explanation for this failure may be the rapid transition (<24 hours) from normal rhythm to third-degree AVB seen in some case reports. Such a rapid transition could only be identified incidentally by weekly fetal echocardiograms.

The pathogenesis of the disease, mediated by the transplacental passage of anti-Ro/SSA antibodies through the neonatal Fc receptor, is not well understood, but is probably due to the inflammatory cascade following the binding of these antibodies to fetal cardiac myocytes.

Extranodal diseases such as dilated cardiomyopathy, valvular regurgitation and endocardial fibroelastosis (EFE) could be associated with AVB. Few data are available on risk stratification based on antibody levels.

One of the major challenges in examining the pathophysiology of CHB is to elucidate the mechanism by which maternal autoantibodies initiate lesions at antigen sites, which are normally intracellular.

One hypothesis is that Ro/La antigens transfer to the surface of cardiomyocytes undergoing normal physiological remodelling, allowing access to the antigens by circulating autoantibodies and triggering subsequent immune responses. Furthermore, in vitro studies have demonstrated that normal fetal cardiocytes are capable of engulfing apoptotic cardiocytes; the formation of immune complexes on phagocytic cardiocytes can impair their clearance by healthy cardiocytes, impeding a function critical to the normal development of the fetal heart. Indeed, histological evaluation of normal fetal hearts shows virtually no apoptotic cells, while the hearts of fetuses that die with CHB show extensive apoptosis. In turn, apoptotic cells lead to infiltration by macrophages, whose subsequent activation causes the release of pro-inflammatory and fibrotic cytokines such as TNFα and thus tissue damage and fibrosis.

Another hypothesis suggests that there is cross-reactivity of Ro antibodies with L-type calcium channels (LTCCs) on the surface of cardiomyocytes, which disrupts calcium homeostasis and produces conduction abnormalities. The LTCC is critical for the generation of action potential in the sinoatrial and atrioventricular nodes, both prone to lesions resulting from neonatal lupus.

Another study demonstrated that pups develop sinus bradycardia and heart block when passively immunized to Ro/La antibodies. Furthermore, over-expression of LTCC could prevent heart block upon exposure to Ro/La antibodies, suggesting that these antibodies negatively affect LTCC function.

Low penetrance of autoimmune CHB in mothers with Ro/La antibodies may indicate protective factors in the fetus. β2-GPI has been shown to bind to apoptotic fetal cardiomyocytes in a dose-dependent manner and prevent opsonization of apoptotic cardiomyocytes by maternal IgG Ro60. Furthermore, cord blood from autoimmune CHB-affected infants showed significantly lower levels of β2-GPI than unaffected infants, suggesting that β2-GPI may be protective for a fetus in a pregnancy exposed to Ro antibodies .

Furthermore, hearts from fetuses that died of autoimmune CHB showed exaggerated apoptosis compared to electively terminated fetal hearts. Apoptosis was accompanied by increased TGF-β immunoreactivity in the extracellular matrix and macrophage infiltration. Increased SMAc staining of transdifferentiating myofibroblasts and increased collagen expression in cardiac fibroblasts have been shown to be consequences of TGF-β activation.

Endocardial fibroelastosis (EFE) deserves special mention as a form of myocardial fibrosis found in 7% of children with autoimmune CHB, although a clear association between the two conditions has not been demonstrated. EFE can lead to end-stage heart failure and subsequent death: a previous study showed that children with EFE had a 51% mortality rate, and in those with concurrent cardiomyopathy that rate rose as high as 100%. EFE can be detected on echocardiograms as areas of irregular echogenicity on the endocardial surfaces of the fetal heart.

Valvular disease is another rare but serious complication of autoimmune CHB, with tensor apparatus dysfunction occurring in 1.6% of cases. Echocardiographic studies show irregular papillary muscle echogenicity, detected between 19-22 weeks, involving the tricuspid and mitral valves. Valvular regurgitation can develop both prenatally and postnatally, from 34 weeks of gestation to 26 weeks after birth. All of the children needed urgent valve surgery.

Dilated cardiomyopathy (DCM) is the other significant, albeit rare, cardiac complication found in children with autoimmune CHB, associated with a high mortality rate. In DCM, the left ventricle is enlarged and weakened, resulting in a decreased ability of the heart to pump blood. DCM can be diagnosed in utero along with CHB, but can also manifest after birth as postnatal DCM. Risk factors for DCM remain unclear. Two distinct types of DCM have been demonstrated: neonatal DCM and late-onset DCM. Hydrops, EFE, and pericardial effusion were all associated with neonatal DCM; factors associated with late-onset DCM were non-European ancestry, pacemaker implantation, and valve regurgitation. Notably, the use of fluorinated steroids had no protective effect against late-onset DCM, and none of the risk factors associated with neonatal DCM were predictive of late-onset DCM.

As previously demonstrated, AV block progresses from "incomplete" block (first degree - AVB I) to "complete" block (third degree - AVB III) and this progression could theoretically be detected by a prolongation of the AV interval (from normal at +3 SD or at >150ms); in the early stages, the detection of alterations in the fetal heart rhythm, through a fetal cardiac Doppler performed at home directly by the patient could allow an early identification of the problem, the rapid access of the patient to the reference Gynecology and Obstetrics Center, where the patient will perform fetal ultrasound with possible confirmation of AV block, and early diagnosis with rapid access to internationally recommended treatment. Treatment of grade I or II AVB with dexamethasone and other therapies may prevent progression to grade III AVB.

Transition from incomplete AV block to grade III AVB has been shown to occur in less than 24 hours, which therefore also appears to be the window of opportunity for effective treatment; this suggests that incomplete AVB can only occasionally be detected by weekly echocardiography. Conversely, frequent (twice daily) home monitoring of fetal heart rhythm (FHR) by mothers can detect second-degree AVB, thus identifying the therapeutic window for treatment success.

Finally, the echocardiogram assessing the mechanical AV interval appears to overestimate the electrical PR interval, with the possibility of detecting the transition from normal rhythm to the echocardiographic equivalent of AVB I, which is not pathological and is transient in some cases.

Some of the factors that increase the risk of developing CHB include a positive family history of CHB in previous pregnancies and high levels of antibodies. The risk increases to 15%-20% for those with a positive family history in a previous pregnancy with CHB. Another high-risk group are patients with high levels of antibodies. In a recent study of pregnancy risk, stratified by anti-Ro/SSA levels, no cases of conduction abnormalities were found in pregnancies with an antibody level below 50 U/mL. Conversely, 8/127 (6%) of fetuses with levels above 50 U/mL developed conduction abnormalities and 3% had CHB.

Several studies show that maternal Ro/SSA antibodies, like all maternal IgG, cross the placenta starting in the early second trimester. Between weeks 17 and 22, the infant has <10% of the maternal IgG level, with levels increasing markedly between weeks 25 and 40. Due to a large increase in umbilical cord blood levels that occurs after week 36 of gestation, preterm infants have lower total IgG levels.

IgG1 appears to be preferentially transported over IgG2, IgG3 and IgG4 by FcRn, with infant IgG1 levels at term delivery nearly double maternal levels. Exposure of the developing fetal AVB to maternal Ro/SSA antibodies leads to local inflammation and, eventually, permanent scarring of the fetal AV node.

Once damaged, the AV node is unable to transmit heart rhythm from the atrium to the ventricle, and the ventricular rate relies on a slow escape mechanism to provide cardiac output. Over the past two decades, physicians have made efforts to identify CHB early and stop its progression. In particular, some groups have tried to monitor changes in the fetal heart that may precede CHB using the fetal echocardiogram.

Once identified, these changes have sometimes been treated with dexamethasone, a corticosteroid that crosses the placenta. However, the results of these screening and treatment efforts have been mixed. Large-scale studies are limited by the rarity of the disease. More recent data indicate that patients taking hydroxychloroquine (HCQ) during pregnancy may have lower rates of CHB in their offspring, suggesting that this drug may prevent CHB.

Because large-scale randomized trials have not been conducted, there is limited clinical data and no official guidelines. Therefore, clinicians are left with some ideas, but limited evidence to clearly support approaches to prevent, predict, or treat CHB.

In a recent consensus document by Clowse et al., for anti-Ro/SSA positive pregnant women followed up in dedicated centres, 80% of 49 experts recommended screening by serial fetal echocardiogram, with the majority of respondents (59%) who suggested starting echocardiograms at week 16 and stopping screening at week 28, even though there was no agreement on which week to stop screening. For women with no history of neonatal lupus, respondents recommend a fetal echocardiogram every other week (44%) or weekly (28%). For women with a previous baby with neonatal lupus, 80% recommend a weekly fetal echocardiogram. To prevent CHB, HCQ was recommended by 67% of respondents and most would start before pregnancy (62%). Respondents were asked for medication guidelines for the treatment of varying degrees of CHB in a 20-week pregnant, anti-Ro and anti-La positive SLE female patient. For first degree, respondents recommended starting dexamethasone (53%) or HCQ (43%). For second degree, respondents recommended starting dexamethasone (88%). For third degree, respondents recommended starting dexamethasone (55%) or IVIg (33%), although 27% would not start any treatment.

Despite the absence of official guidelines, in fact, many physicians with a focus on pregnancy and rheumatic diseases have developed similar models in the screening, prevention and treatment of CHB, so much so that monitoring the fetal heart rate with fetal heart Doppler at domicile, to be performed bis or tris in die, represents a consolidated approach of "good clinical practice".

Cardiac manifestations do not occur randomly, but rather occur over a fairly well-defined period, between 18 and 26 weeks, allowing clinicians to focus more closely on the surveillance period.

Hypothesis under study Progression from normal sinus rhythm to complete heart block can be rapid, occurring in a week or less. High-dose steroid or high-dose gamma globulin therapy used a few days after detection of complete block has yielded controversial results. However, it is possible that in the early hours there is a window of opportunity during which immunosuppressive therapy can reverse some very initial damage.

Detection of heart block is usually performed with a surface ECG, but while the fetus is in the uterine cavity this method is not applicable. The normal fetal heart rate is 100-130 bpm. In the presence of advanced conduction blocks, not all atrial contractions are transmitted to the ventricles, and the recorded frequency (which is the ventricular one) drops by a lot, reaching 70-80 bpm or even lower values; such low frequencies (for the fetus) often correspond to the appearance of extrasystoles or in any case of irregular heartbeats, given that only some atrial contractions are transmitted to the ventricles. A heart-frequency monitor, highlighting bradycardia and/or irregularities in the heartbeat, can give valuable indications to suggest the appearance of a heart block very early. However, this blockage will then be precisely detected by a fetal echocardiogram performed within a few hours on the basis of the suspicion highlighted with the heart rate monitor. The hypothesis is that in such an early stage there is a window of opportunity to promptly use the available therapies.

The heart rate monitor therefore raises the suspicion, and the subsequent complete fetal ultrasound will confirm or not the diagnosis.

If fetal heart rhythm surveillance could be shown to detect a medically reversible disease that, if untreated, would progress to lifelong cardiac pacing, with its many associated comorbidities, applying such a protocol in pregnant women anti-Ro/SSA positive could become standard practice as already happens in other countries.

Similarly, universal prenatal screening of all pregnant women for the presence of anti-Ro/SSA antibodies would be warranted.

Previously, Cuneo et al. demonstrated the feasibility of monitoring fetal heart rate with a home-use Doppler device. In this project, anti-Ro/SSA-positive pregnant women monitored fetal heart rate and rhythm twice daily in the home setting and underwent a fetal echocardiogram if the fetal heart rhythm was irregular. The first experience was subsequently extended to 273 anti-Ro/SSA positive pregnancies, both monitored by both echocardiography and home fetal heart rate monitoring, with encouraging results.

From a more recent investigation, the same group concluded that the diagnostic threshold for grade I BAV depends on gestational age.

Also, Brucato et al. previously published a case report of a 31-year-old woman with SLE and positive serology for anti-Ro/SSA antibodies, who underwent home monitoring of fetal heart rate with a Doppler device. At the 26th week of pregnancy, during the monitoring, the mother found an arrhythmia. A fetal echocardiogram was performed within a few hours, which did not document rhythm abnormalities, for which the patient continued with home monitoring.

Purpose of the study The aim of the present study is to evaluate the incidence of fetal BAV of various degrees in pregnant patients carrying anti-SSA autoantibodies, by monitoring the fetal heart rate performed every eight hours at home after instruction on the use of the device. If this monitoring detects bradycardia or fetal heartbeat irregularities, a complete fetal ultrasound examination will be quickly performed subsequently to confirm or not the suspicion posed by the monitoring performed at home. This study will therefore evaluate the incidence of this pathology of the fetal rhythm in patients with such autoantibody positivity and the same patients will then have the possibility of accessing the treatments for this fetal pathology recommended at an international level.

In addition to the estimated incidence of cases of BAV in fetuses of pregnant women with anti Ro/SSA antibodies, through this study investigators will be able to evaluate whether a very early treatment can improve the final outcome.

ELIGIBILITY:
Inclusion Criteria:

* All patients over the age of 18 will be enrolled in the study, who will sign the informed consent for participation in the study, characterized by the positivity of autoantibodies against Ro/SSA who will become pregnant during the enrollment period in the enrolling centres.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: All patients over the age of 18 characterized by the positivity of autoantibodies against Ro/SSA who will become pregnant during the enrollment period in the enrolling centres.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-04-14 (Actual); Primary Completion 2025-04-14 (Estimated); Study Completion 2026-04-14 (Estimated)

PRIMARY OUTCOMES:
Incidence of fetal atrio-ventricular block evaluated as percentage of patients experiencing a fetal atrio-ventricular block. | 8 months
  Estimation of the incidence of fetal heart disease in pregnant patients with positive SSA autoantibodies

SECONDARY OUTCOMES:
Home fetal heart rate monitoring reliability: percentage of patients reporting alterations of fetal heart rhythm detected by the hand-held fetal heart rate doppler. | 5 months
  Estimate of the reliability of home monitoring of fetal heart rate with fetal Doppler device and its possible usefulness in the early diagnosis of fetal heart rhythm disturbances.
  Data will be reported as percentage of patients reporting alterations of fetal heart rhythm detected by the hand-held fetal heart rate doppler and percentage of eventual confirmations of fetal heart rhythm alteration by the use of heart fetal ultrasound examination performed within 8 hours of fetal heart rhythm alteration detected by home monitoring.
Therapies' outcomes: percentage of patients where fetal atrio-ventricular block will be reverted by the use of individualized therapies. | 8 months
  Evaluation of the results of rapidly prepared therapy in cases of ultrasound confirmation of fetal heart rhythm disturbances reported as the percentage of patients where the therapy proved successful in reverting the atrio-ventricular block.
Pregnancy outcome other than atrio-ventricular block reported as percentage of newborns presenting other symptoms of neonatal lupus, subgroup: hepatologic manifestations. | 8 months
  Evaluation, expressed as percentage of total newborns, of pregnancy outcomes other than atrioventricular block: hepatological manifestations.
Pregnancy outcome other than atrio-ventricular block. Percentage of newborns presenting other symptoms of neonatal lupus, subgroup: haematologic manifestations. | 8 months
  Evaluation, expressed as percentage of total newborns, of pregnancy outcomes other than atrioventricular block: haematological manifestations.
Pregnancy outcome other than atrio-ventricular block. Percentage of newborns presenting other symptoms of neonatal lupus, subgroup: skin conditions. | 8 months
  Evaluation, expressed as percentage of total newborns, of pregnancy outcomes other than atrioventricular block: skin conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Luca Brucato, Prof, Principal Investigator — ASST Fatebenefratelli, Milano, Italy
Locations (1):
- ASST Fatebenefratelli e Sacco, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wilhelm BJ, Thone M, El-Scheich T, Livert D, Angelico R, Osswald B. Complications and Risk Assessment of 25 Years in Pediatric Pacing. Ann Thorac Surg. 2015 Jul;100(1):147-53. doi: 10.1016/j.athoracsur.2014.12.098. Epub 2015 May 14. PMID 25980596
- [Result] Wainwright B, Bhan R, Trad C, Cohen R, Saxena A, Buyon J, Izmirly P. Autoimmune-mediated congenital heart block. Best Pract Res Clin Obstet Gynaecol. 2020 Apr;64:41-51. doi: 10.1016/j.bpobgyn.2019.09.001. Epub 2019 Oct 8. PMID 31685414
- [Result] Brucato A, Frassi M, Franceschini F, Cimaz R, Faden D, Pisoni MP, Muscara M, Vignati G, Stramba-Badiale M, Catelli L, Lojacono A, Cavazzana I, Ghirardello A, Vescovi F, Gambari PF, Doria A, Meroni PL, Tincani A. Risk of congenital complete heart block in newborns of mothers with anti-Ro/SSA antibodies detected by counterimmunoelectrophoresis: a prospective study of 100 women. Arthritis Rheum. 2001 Aug;44(8):1832-5. doi: 10.1002/1529-0131(200108)44:83.0.CO;2-C. PMID 11508435
- [Result] Fredi M, Andreoli L, Bacco B, Bertero T, Bortoluzzi A, Breda S, Cappa V, Ceccarelli F, Cimaz R, De Vita S, Di Poi E, Elefante E, Franceschini F, Gerosa M, Govoni M, Hoxha A, Lojacono A, Marozio L, Mathieu A, Meroni PL, Minniti A, Mosca M, Muscara M, Padovan M, Piga M, Priori R, Ramoni V, Ruffatti A, Tani C, Tonello M, Trespidi L, Zatti S, Calza S, Tincani A, Brucato A. First Report of the Italian Registry on Immune-Mediated Congenital Heart Block (Lu.Ne Registry). Front Cardiovasc Med. 2019 Feb 28;6:11. doi: 10.3389/fcvm.2019.00011. eCollection 2019. PMID 30873413
- [Result] Brucato A, Tincani A, Fredi M, Breda S, Ramoni V, Morel N, Costedoat-Chalumeau N. Should we treat congenital heart block with fluorinated corticosteroids? Autoimmun Rev. 2017 Nov;16(11):1115-1118. doi: 10.1016/j.autrev.2017.09.005. Epub 2017 Sep 9. No abstract available. PMID 28899797
- [Result] Friedman DM, Kim MY, Copel JA, Davis C, Phoon CK, Glickstein JS, Buyon JP; PRIDE Investigators. Utility of cardiac monitoring in fetuses at risk for congenital heart block: the PR Interval and Dexamethasone Evaluation (PRIDE) prospective study. Circulation. 2008 Jan 29;117(4):485-93. doi: 10.1161/CIRCULATIONAHA.107.707661. Epub 2008 Jan 14. PMID 18195175
- [Result] Sonesson SE, Ambrosi A, Wahren-Herlenius M. Benefits of fetal echocardiographic surveillance in pregnancies at risk of congenital heart block: single-center study of 212 anti-Ro52-positive pregnancies. Ultrasound Obstet Gynecol. 2019 Jul;54(1):87-95. doi: 10.1002/uog.20214. Epub 2019 Jun 7. PMID 30620419
- [Result] Cuneo BF, Bitant S, Strasburger JF, Kaizer AM, Wakai RT. Assessment of atrioventricular conduction by echocardiography and magnetocardiography in normal and anti-Ro/SSA-antibody-positive pregnancies. Ultrasound Obstet Gynecol. 2019 Nov;54(5):625-633. doi: 10.1002/uog.20245. PMID 30784137
- [Result] Izmirly PM, Buyon JP, Saxena A. Neonatal lupus: advances in understanding pathogenesis and identifying treatments of cardiac disease. Curr Opin Rheumatol. 2012 Sep;24(5):466-72. doi: 10.1097/BOR.0b013e328356226b. PMID 22832822
- [Result] Miner JJ, Kim AH. Cardiac manifestations of systemic lupus erythematosus. Rheum Dis Clin North Am. 2014 Feb;40(1):51-60. doi: 10.1016/j.rdc.2013.10.003. PMID 24268009
- [Result] Jaeggi E, Laskin C, Hamilton R, Kingdom J, Silverman E. The importance of the level of maternal anti-Ro/SSA antibodies as a prognostic marker of the development of cardiac neonatal lupus erythematosus a prospective study of 186 antibody-exposed fetuses and infants. J Am Coll Cardiol. 2010 Jun 15;55(24):2778-84. doi: 10.1016/j.jacc.2010.02.042. PMID 20538173
- [Result] Buyon JP, Clancy RM. Neonatal lupus: review of proposed pathogenesis and clinical data from the US-based Research Registry for Neonatal Lupus. Autoimmunity. 2003 Feb;36(1):41-50. doi: 10.1080/0891693031000067340. PMID 12765470
- [Result] Brucato A, Previtali E, Ramoni V, Ghidoni S. Arrhythmias presenting in neonatal lupus. Scand J Immunol. 2010 Sep;72(3):198-204. doi: 10.1111/j.1365-3083.2010.02441.x. PMID 20696016
- [Result] Eftekhari P, Roegel JC, Lezoualc'h F, Fischmeister R, Imbs JL, Hoebeke J. Induction of neonatal lupus in pups of mice immunized with synthetic peptides derived from amino acid sequences of the serotoninergic 5-HT4 receptor. Eur J Immunol. 2001 Feb;31(2):573-9. doi: 10.1002/1521-4141(200102)31:23.0.co;2-9. PMID 11180122
- [Result] Reed JH, Clancy RM, Purcell AW, Kim MY, Gordon TP, Buyon JP. beta2-glycoprotein I and protection from anti-SSA/Ro60-associated cardiac manifestations of neonatal lupus. J Immunol. 2011 Jul 1;187(1):520-6. doi: 10.4049/jimmunol.1100122. Epub 2011 May 20. PMID 21602492
- [Result] Clancy RM, Buyon JP. Autoimmune-associated congenital heart block: dissecting the cascade from immunologic insult to relentless fibrosis. Anat Rec A Discov Mol Cell Evol Biol. 2004 Oct;280(2):1027-35. doi: 10.1002/ar.a.20072. PMID 15368347
- [Result] Tincani A, Rebaioli CB, Taglietti M, Shoenfeld Y. Heart involvement in systemic lupus erythematosus, anti-phospholipid syndrome and neonatal lupus. Rheumatology (Oxford). 2006 Oct;45 Suppl 4:iv8-13. doi: 10.1093/rheumatology/kel308. PMID 16980725
- [Result] Morel N, Levesque K, Maltret A, Baron G, Hamidou M, Orquevaux P, Piette JC, Barriere F, Le Bidois J, Fermont L, Fain O, Theulin A, Sassolas F, Hauet Q, Guettrot-Imbert G, Georgin-Lavialle S, Deligny C, Hachulla E, Mouthon L, Le Jeunne C, Ravaud P, Le Mercier D, Romefort B, Villain E, Bonnet D, Costedoat-Chalumeau N; "Lupus neonatal" group. Incidence, risk factors, and mortality of neonatal and late-onset dilated cardiomyopathy associated with cardiac neonatal lupus. Int J Cardiol. 2017 Dec 1;248:263-269. doi: 10.1016/j.ijcard.2017.07.100. Epub 2017 Aug 7. PMID 28843719
- [Result] Izmirly PM, Saxena A, Kim MY, Wang D, Sahl SK, Llanos C, Friedman D, Buyon JP. Maternal and fetal factors associated with mortality and morbidity in a multi-racial/ethnic registry of anti-SSA/Ro-associated cardiac neonatal lupus. Circulation. 2011 Nov 1;124(18):1927-35. doi: 10.1161/CIRCULATIONAHA.111.033894. Epub 2011 Oct 3. PMID 21969015
- [Result] Cuneo BF, Sonesson SE, Levasseur S, Moon-Grady AJ, Krishnan A, Donofrio MT, Raboisson MJ, Hornberger LK, Van Eerden P, Sinkovskaya E, Abuhamad A, Arya B, Szwast A, Gardiner H, Jacobs K, Freire G, Howley L, Lam A, Kaizer AM, Benson DW, Jaeggi E. Home Monitoring for Fetal Heart Rhythm During Anti-Ro Pregnancies. J Am Coll Cardiol. 2018 Oct 16;72(16):1940-1951. doi: 10.1016/j.jacc.2018.07.076. PMID 30309472
- [Result] Feki S, Turki A, Frikha F, Hachicha H, Walha L, Gargouri A, Bahloul Z, Masmoudi H. [Neonatal lupus and maternofetal transmission of anti-SSA/Ro and anti-SSB/La antibodies]. Arch Pediatr. 2015 Feb;22(2):154-9. doi: 10.1016/j.arcped.2014.10.020. Epub 2014 Nov 13. French. PMID 25440767
- [Result] Ciobanu AM, Dumitru AE, Gica N, Botezatu R, Peltecu G, Panaitescu AM. Benefits and Risks of IgG Transplacental Transfer. Diagnostics (Basel). 2020 Aug 12;10(8):583. doi: 10.3390/diagnostics10080583. PMID 32806663
- [Result] Izmirly PM, Costedoat-Chalumeau N, Pisoni CN, Khamashta MA, Kim MY, Saxena A, Friedman D, Llanos C, Piette JC, Buyon JP. Maternal use of hydroxychloroquine is associated with a reduced risk of recurrent anti-SSA/Ro-antibody-associated cardiac manifestations of neonatal lupus. Circulation. 2012 Jul 3;126(1):76-82. doi: 10.1161/CIRCULATIONAHA.111.089268. Epub 2012 May 24. PMID 22626746
- [Result] Clowse MEB, Eudy AM, Kiernan E, Williams MR, Bermas B, Chakravarty E, Sammaritano LR, Chambers CD, Buyon J. The prevention, screening and treatment of congenital heart block from neonatal lupus: a survey of provider practices. Rheumatology (Oxford). 2018 Jul 1;57(suppl_5):v9-v17. doi: 10.1093/rheumatology/key141. PMID 30137589
- [Result] Milazzo R, Ligato E, Laoreti A, Ferri G, Basili L, Serati L, Brucato A, Cetin I. Home fetal heart rate monitoring in anti Ro/SSA positive pregnancies: Literature review and case report. Eur J Obstet Gynecol Reprod Biol. 2021 Apr;259:1-6. doi: 10.1016/j.ejogrb.2021.01.031. Epub 2021 Jan 28. PMID 33556767
- [Result] Sunderji S, Peyvandi S, Jaeggi E, Szwast A, Ryan G, Tessier F, Siddiqui S, Cuneo B, Sheth S, Treadwell M, Frommelt M, Turan S, Copel J, Emery S, Rand L, Moon-Grady AJ; North American Fetal Therapy Network (NAFTNet). NAFTNet retrospective report on the treatment of anti-Ro/SSA mediated fetal heart block with dexamethasone. J Matern Fetal Neonatal Med. 2022 Dec;35(25):9263-9270. doi: 10.1080/14767058.2022.2025536. Epub 2022 Jan 11. PMID 35014577